CLINICAL TRIAL: NCT05476705
Title: Right Place, Right Practitioner, Right Time: Development of Emergency Department Triage to Support the Identification and Management of Drug Related Problems
Brief Title: Identifying Drug-related Problems at ED Triage (DRP-EDiT) V1
Acronym: DRP-EDiT
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Anglia Ruskin University (Other)
Collaborators: Pharmacy Research UK (Unknown); University of Manchester (Other); Ashford and St. Peter's Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: IRAS 307523
Record Dates: First submitted 2022-07-22; First posted 2022-07-27 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2022-07

CONDITIONS: Medication Administered in Error; Medication Adverse Effects; Medication Reaction
Keywords: Drug-related problems; Emergency department; Triage; Identification; Management; Pharmacists
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions; Emergencies

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Up to a third of patients who visit emergency departments (EDs) do so because they have an issue with medicines prescribed by their doctor or purchased over the counter. For example, some patients might experience side effects (e.g., sickness), whereas others may feel their prescribed medicine is not working and want an alternative. While some patients who visit EDs know they have a problem with their medication, some are not aware. Furthermore, drug-related problems (DRPs) may not be identified by ED triage systems which are used to sort patients' priority for treatment. The currently used system in the UK (Manchester Triage System) mentions drugs infrequently and does not support the identification of the most common DRPs. For this project, DRPs include medication errors, adverse drug events, and adverse drug reactions. This project aims to revise the triage system to support the discovery of patients' medication problems when they are triaged by a nurse upon arrival to the ED.

After identification, problems with a patient's medication should be dealt with by the healthcare professional who is most appropriate to manage that particular issue. For example, a patient who has been prescribed a new medicine but already takes 20 medicines will likely benefit from a review by a pharmacist in the ED. This project will aim to support the management of patients who might benefit from care provided by pharmacists by providing them with this care.

As well as ensuring medication problems are identified at triage, and that pharmacists are involved in helping to deal with those problems, this project will also try to understand how we can investigate how pharmacists actually make a difference to the care of ED patients.

A multi-step approach (Stages A-F) is proposed to answer the question "How can patient DRPs be identified, triaged and managed in the ED?" In summary, the steps include: STAGE A, a systematic review and scoping survey; STAGE B, researcher visits to ED sites to shadow ED staff; STAGE C, Interviews with healthcare professionals (including those shadowed in STAGE B) to validate findings of site visits and explore topics in more depth; STAGE D, developing additional drug-related content for the Manchester Triage System; STAGE E, involving a panel of experts in a RAND appropriateness method to rate the content developed in STAGE D; STAGE F, testing the revised triage system for a future pilot study involving interviews with staff visited in STAGE B.

ELIGIBILITY:
Inclusion Criteria: The following groups will be included in various stages of the project

* STAGE A: ED clinicians at UK-wide NHS trusts
* STAGE B: ED staff from 8 NHS sites across the UK
* STAGE C: ED staff from 8 NHS sites across the UK
* STAGE E: Clinicians and academics with expertise in Emergency Care and/or ED Triage
* STAGE F: ED staff from 8 NHS sites across the UK

Exclusion Criteria:

* Those who do not consent or who are unable to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Hospital Emergency Department staff and clinicians and academics with expertise in Emergency Care and/or ED Triage
Sampling Method: Non-Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2023-04 (Estimated); Primary Completion 2023-09 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Suitability of a revised Manchester Triage System (MTS) | 13 months (the revised MTS will be an output from the analysis of data collected months 1 - 13)
  The suitability of a revised MTS to support identification and management of drug-related problems in the Emergency Department

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Greenwood, Principal Investigator — Anglia Ruskin University